CLINICAL TRIAL: NCT04779242
Title: A Phase 3b Randomized, Double-Blind, Multi-Center Study to Compare the Safety and Efficacy of Omadacycline IV/PO to Moxifloxacin IV/PO for Treating Adult Subjects With Community-Acquired Bacterial Pneumonia (CABP)
Brief Title: Omadacycline vs. Moxifloxacin for the Treatment of Community-Acquired Bacterial Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTK0796-CABP-19302
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Community-acquired Pneumonia; Bacterial Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia, Bacterial | interventions — omadacycline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omadacycline (Experimental): Omadacycline 100 mg IV; Omadacycline 300 mg PO (2 x 150 mg tablets); QD Dosing; 7-10 day duration.
  Interventions: Drug: Omadacycline
- Moxifloxacin (Active Comparator): Moxifloxacin 400 mg IV; Moxifloxacin 400 mg tablets; QD Dosing; 7-10 day duration
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Omadacycline — IV for injection, oral tablets
  Other Names: NUZYRA
  Arms: Omadacycline
Drug: Moxifloxacin — IV solution, oral tablets
  Other Names: Avelox
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of omadacycline as compared to moxifloxacin in the treatment of adults with community-acquired bacterial pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age 18 or older who have signed the informed consent form
* Must have a qualifying community-acquired bacterial pneumonia
* Subjects must not be pregnant or nursing at the time of enrollment
* Must agree to a reliable method of birth control during the study and for 30 days following the last dose of study drug

Exclusion Criteria:

* Known or suspected hospital-acquired pneumonia
* Confirmed or suspected SARS-CoV-2 infection
* Evidence of significant immunological disease
* Has a life expectancy of less than or equal to 3 months or any concomitant condition that is likely to interfere with evaluation of the response of the infection under study, determination of AEs, or completion of the expected course of treatment
* Has a history of contraindications, hypersensitivity, or allergic reaction to any tetracycline or fluoroquinolone antibiotic
* Has received an investigational drug within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Manley, Study Director — Paratek Pharmaceuticals Inc
Locations (55):
- Bulgaria (12):
  - Site 210, Gabrovo
  - Site 213, Lom
  - Site 208, Pernik
  - Site 201, Pleven
  - Site 206, Rousse
  - Site 207, Sliven
  - Site 202, Sofia
  - Site 204, Sofia
  - Site 205, Sofia
  - Site 209, Sofia
  - Site 212, Vidin
  - Site 211, Vratsa
- Croatia (4):
  - Site 302, Split
  - Site 301, Zagreb
  - Site 303, Zagreb
  - Site 304, Zagreb
- Georgia (7):
  - Site 401, Tbilisi
  - Site 402, Tbilisi
  - Site 403, Tbilisi
  - Site 404, Tbilisi
  - Site 405, Tbilisi
  - Site 406, Tbilisi
  - Site 407, Tbilisi
- Hungary (5):
  - Site 802, Balassagyarmat
  - Site 801, Budapest
  - Site 803, Debrecen
  - Site 804, Kistarcsa
  - Site 805, Törökbálint
- Poland (4):
  - Site 901, Chrzanów
  - Site 904, Krakow
  - Site 902, Oświęcim
  - Site 903, Łęczna
- Russia (5):
  - Site 506, Moscow
  - Site 510, Moscow
  - Site 507, Saint Petersburg
  - Site 508, Saint Petersburg
  - Site 509, Saint Petersburg
- Serbia (8):
  - Site 703, Belgrade
  - Site 704, Belgrade
  - Site 705, Belgrade
  - Site 707, Belgrade
  - Site708, Belgrade
  - Site 706, Kamenitz
  - Site 701, Kragujevac
  - Site 702, Niš
- Ukraine (10):
  - Site 606, Dnipro
  - Site 602, Kharkiv
  - Site 604, Kharkiv
  - Site 611, Kharkiv
  - Site 603, Kyiv
  - Site 605, Kyiv
  - Site 607, Kyiv
  - Site 609, Kyiv
  - Site 608, Zaporizhia
  - Site 610, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, double-blind, active comparator-controlled study comparing Omadacycline and Moxifloxacin with participants with Community-Acquired Bacterial Pneumonia (CABP). The randomization was stratified by Pneumonia Outcomes Research Team (PORT) Risk Class (III or IV), and receipt of an allowed antibacterial therapy in the 72 hours prior to study treatment.
Pre-assignment Details: A total of 670 participants were enrolled in approximately 75 sites globally.
Groups:
- Omadacycline: Participants received Omadacycline 200 milligrams (mg) intravenously (IV) once daily or 100 mg IV twice daily on Day 1 and 100 mg IV on Day 2 and 100 mg IV or 300 mg tablets orally once daily from Day 3 through Day 10.
- Moxifloxacin: Participants received Moxifloxacin 400 mg IV on Day 1 and Day 2, and 400 mg IV or as oral tablets from Day 3 through Day 10.
Period: Overall Study
Arm/Group | Omadacycline | Moxifloxacin
Started | 336 | 334
Completed | 308 | 306
Not Completed | 28 | 28
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 7 | 9
Not completed — Death | 6 | 6
Not completed — COVID-19 related reasons | 2 | 1
Not completed — Unavailability for post therapy evaluation Visit | 8 | 4
Not completed — Martial Law in Ukraine | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to Treat (ITT) population consisted of all randomized participants regardless of whether or not the participant received test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | Omadacycline | Moxifloxacin | Total
Number analyzed (Participants) | 336 | 334 | 670
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (14.41) | 62.2 (15.42) | 62.8 (14.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 166 | 324
  Male | 178 | 168 | 346
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 332 | 330 | 662
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 335 | 333 | 668
  Asian | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Early Clinical Response at the Early Clinical Response (ECR) Visit
Description: Early clinical response is defined as clinical success, categorized by survival with improvement of at least 1 level compared to Baseline in at least 2CABP symptoms (cough, sputum production, pleuritic chest pain, and dyspnea) with no worsening in CABP symptoms. Response is determined programmatically using investigator's assessment of the CABP symptoms. The severity of the participant's CABP symptoms was evaluated on a 4-point scale (absent, mild, moderate, or severe) based upon the CABP Subject Symptom Severity Guidance Framework for Investigator Assessment. An indeterminate response is defined as one that could not be adequately inferred because the participant was not assessed because they withdrew consent, or other specified reason. Clinical failure is defined as no improvement by at least 1 level in 2CABP symptoms, worsening of CABP symptom, alternative antibacterial treatment for CABP, discontinuation due to adverse event requiring alternative antibacterial treatment, or death
Time Frame: 72 to 120 hours after the first dose of test article
Population: ITT population
Measure: Number; unit: Percentage of participants
Groups:
- Omadacycline: Participants received Omadacycline 200 mg intravenously (IV) once daily or 100 mg IV twice daily on Day 1 and 100 mg IV on Day 2 and 100 mg IV or 300 mg tablets orally once daily from Day 3 through Day 10.
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 336 | 334
Percentage of participants
  Clinical Success | 89.6 | 87.7
  Clinical Failure | 8.6 | 9.3
  Indeterminate | 1.8 | 3.0
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Other — Difference was observed difference in early clinical success rate between the omadacycline and moxifloxacin groups; Percentage difference = 1.9, 95% CI 2-sided [-3.0 to 6.8] — 95% CI is constructed based on the Miettinen and Nurminen method without stratification

2. Secondary Outcome: Percentage of Participants With Investigator Assessment of Clinical Response at the Post Therapy Evaluation (PTE) Visit
Description: At the PTE Visit, the investigator indicates one of the following outcomes relating to the primary infection under study: Clinical Success: survival after completion of a test article regimen without receiving any systemic antibacterial therapy other than test article, resolution of signs/symptoms of the infection present at Screening with no new symptoms/complications attributable to CABP and no need for further antibacterial therapy. Clinical Failure: alternative antibacterial treatment for CABP was required prior to the PTE Visit related to either (a) progression/development of new CABP symptoms or (b) development of infectious complications of CABP. Other reasons for clinical failure: participant received antibiotics that may have been effective for the infection under study for a different infection from the one under study; death prior to the PTE Visit. Indeterminate: the clinical response to test article could not be adequately inferred.
Time Frame: 5 to 10 days after the last dose of test article
Population: ITT Population
Measure: Number; unit: Percentage of participants
Groups:
- Omadacycline: Participants received Omadacycline 200 mg intravenously once daily or 100 mg IV twice daily on Day 1 and 100 mg IV on Day 2 and 100 mg IV or 300 mg tablets orally once daily from Day 3 through Day 10.
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 336 | 334
Percentage of participants
  Clinical Success | 86 | 87.7
  Clinical Failure | 8.0 | 6.6
  Indeterminate | 6.0 | 5.7
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Other — Difference was observed difference in overall clinical success rate at PTE between the omadacycline and moxifloxacin groups; Percentage difference = -1.7, 95% CI 2-sided [-6.9 to 3.4] — 95% CI is constructed based on the Miettinen and Nurminen method without stratification

3. Secondary Outcome: Percentage of Participants With the Indicated Investigator Assessment of Clinical Response in the Clinically Evaluable-Post Therapy Evaluation (CE-PTE) Population at the PTE Visit
Description: as for outcome 2
Time Frame: 5 to 10 days after the last dose of test article
Population: CE-PTE Population consisted of all ITT participants who received test article, have a qualifying Community-Acquired Bacterial Pneumonia (CABP), an assessment of outcome, and meet all other evaluability criteria.
Measure: Number; unit: Percentage of participants
Groups:
- Omadacycline: Participants received Omadacycline 200 mg IV once or 100 mg IV twice on Day 1 and 100 mg IV on Day 2, and 100 mg IV or 300 mg tablets orally once daily from Day 3 to 10.
Arm/Group | Omadacycline | Moxifloxacin
Number analyzed (Participants) | 273 | 271
Percentage of participants
  Clinical Success | 94.1 | 95.9
  Clinical Failure | 5.9 | 4.1
  Indeterminate | 0 | 0
Statistical Analysis 1: Comparison: Omadacycline vs Moxifloxacin; Test type: Other — [test comment as in outcome 2, analysis 1]; Percentage difference = -1.8, 95% CI 2-sided [-5.7 to 2.0] — 95% CI is constructed based on the Miettinen and Nurminen method without stratification

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the from the first dose of study drug up to the time of the final Follow-up assessment (up to 30 to 37 days after the start of the first infusion of test article)
Arm/Group | Omadacycline | Moxifloxacin
All-Cause Mortality (participants affected / at risk) | 6/336 | 6/332
Serious Adverse Events (participants affected / at risk) | 17/336 | 15/332
Other Adverse Events (participants affected / at risk) | 32/336 | 36/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=336) | Moxifloxacin (N=332)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
COVID-19 (Infections and infestations) | 1 | 2
Infectious pleural effusion (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Pyoderma streptococcal (Infections and infestations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omadacycline (N=336) | Moxifloxacin (N=332)
COVID-19 (Infections and infestations) | 11 | 4
Aspartate aminotransferase increased (Investigations) | 7 | 0
Headache (Nervous system disorders) | 12 | 15
Diarrhoea (Gastrointestinal disorders) | 0 | 10
Insomnia (Psychiatric disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04779242/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT04779242/SAP_001.pdf